CLINICAL TRIAL: NCT06972355
Title: Efficacy of Treadmill Walking With Hidden Vision for Rehabilitation in the Subacute Phase of Stroke, Randomized Controlled Trial
Brief Title: Efficacy of Treadmill Walking With Hidden Vision for Rehabilitation in the Subacute Phase of Stroke
Acronym: MAVREEC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Régional Metz-Thionville (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2025-01-CHRMT
Record Dates: First submitted 2025-04-25; First posted 2025-05-15 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Subacute Stroke
Keywords: Stroke; Gait; Treadmill; Double task; Proprioception; Postural balance
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hidden Eyes (Experimental): Treadmill walking training with body weight reduced and eyes hidden
  Interventions: Procedure: Hiding the eyes
- Open Eyes (No Intervention): Treadmill walking training with reduced body weight and open eyes.

INTERVENTIONS:
Procedure: Hiding the eyes — Patients will participate in walking rehabilitation sessions on a treadmill supported by a Lite Gait® harness. All treadmill sessions are consistent with regular rehabilitation sessions. A typical treadmill walking session will take place 3 times a week for 6 weeks, lasting 20 minutes. During the first minute, the speed of the treadmill is gradually increased until a comfortable speed is reached. From then on, the mask will be placed over the patient's eyes for 18 minutes at a constant, i.e. comfortable, speed. The last minute will be devoted to gradually decreasing the treadmill speed until it stops, and will also be performed without the mask.
  Arms: Hidden Eyes

SUMMARY:
Objective: The aim of this study is to compare the efficiency of vision-obscured versus vision-retained treadmill gait training in subacute post-stroke patients.

Methodology: Thirty-six patients with stroke (ischemic or hemorrhagic) less than six months old will be included and randomized into two parallel groups. The experimental group will undergo treadmill gait training using an opaque mask, combined with body weight reduction (Lite Gait® harness). The control group will follow the same walking protocol, but with their eyes open. Each session will last 20 minutes, integrated into one hour of rehabilitation, at a rate of three sessions per week for six weeks. Assessment will include single- and double-task walking speed, balance parameters and proprioception.

Expected results: The hypothesis is that visual deprivation will stimulate the proprioceptive and vestibular systems to a greater extent, resulting in benefits for postural balance, walking and proprioception. The main hypothesis will be the improvement in the difference between single-task and double-task walking speed. Analyses will be conducted on an intention-to-treat basis, using statistical tests adapted to the nature of the variables.

Conclusion: This study could highlight the value of temporary visual suppression as a therapeutic lever in stroke rehabilitation.

DETAILED DESCRIPTION:
Background: Gait rehabilitation for stroke patients is a major issue in post-stroke functional recovery. The impact of vision on walking and balance is well documented, however, visuo-dependence (the dependence on vision for spatial orientation and balance control) is often neglected in current rehabilitation programs. Programs dealing with visuo-dependence mainly target pediatric, geriatric or chronic stroke populations, but their use and study remain limited in the literature. Moreover, these programs have never been studied in the context of the sub-acute phase of stroke. The issue of visuo-dependence is particularly relevant in this phase, as it occurs at a time when brain plasticity is still possible and appropriate rehabilitation strategies are needed.

Aims

The primary aim of this study is to evaluate the effects of treadmill walking training with vision suppression (eyes closed) on double-task walking speed.

Secondary objectives are to study balance parameters, including lateral variance of the center of pressure (with eyes open and closed), area covered by the center of pressure (eyes open and closed), Romberg quotient and MCTSIB score. Gait parameters such as 10-meter test speed (10MWT), mean step duration, symmetry and cycle length variability will also be studied. Finally, proprioception parameters will be assessed using the JPS test.

The primary hypothesis is that the absence of vision significantly improves the difference in walking speed between single-task and double-task walking. The secondary hypothesis is that this absence of vision would also improve proprioception parameters, gait quality and balance, by forcing increased activation of the other senses (proprioception, vestibular system), thus leading to somatosensory compensation.

Methodology

This randomized, controlled study will involve sub-acute stroke patients (< 6 months), aged over 18, with deficits in walking, balance and proprioception. Participants will be randomly divided into two groups: an experimental group receiving gait training with eyes closed, and a control group practicing training with eyes open. Each participant will follow a rehabilitation program of 20 minutes of treadmill walking, three times a week, as part of physical therapy sessions lasting one hour a day, 5 times a week. Inclusion criteria included the ability to walk for 20 minutes on a treadmill with suspension and to walk 10 metres in the corridor, with or without technical aids. Exclusion criteria included severe associated pathologies and major cognitive impairment.

Conclusion and clinical implications : This study is innovative in that it explores the effects of vision suppression on gait and balance rehabilitation, specifically in sub-acute stroke patients, a population often neglected in existing research. The results could offer new perspectives for post-stroke rehabilitation, focusing on sensory compensation via proprioception and other senses. This approach could ultimately improve patients' quality of life and autonomy, by reducing their dependence on vision and optimizing their motor rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age or older,
2. With a confirmed diagnosis of ischemic or hemorrhagic stroke in sub-acute phase (stroke less than 6 months old),
3. With NIHSS scores between 1 and 15 and MoCA scores between 18 and 30
4. With a physiotherapy prescription for post Stroke rehabilitation
5. Able to walk for 20 min on a treadmill with weight reduction with pauses, able to maintain bipodal balance, able to maintain bipodal balance with eyes open and closed for 30 seconds,
6. Having expressed free, informed and written consent
7. Affiliated with a social security scheme.

Exclusion Criteria:

1. Patients weighing over 200 kg (maximum weight permitted for use of the Lite Gait ®),
2. Patients with impaired vision:

   1. Best corrected visual acuity below 5/10 on patient examination
   2. Homonymous lateral hemianopia, quadranopia.
3. Inability to physically participate in intensive rehabilitation due to severe, unstabilized and comorbidities (heart, lung, kidney disease or diabetes), severe psychiatric disorders cancer active or under treatment.
4. Patients participating in other interventional research,
5. Pregnant or breast-feeding women,
6. Patients under guardianship.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2025-06-04 (Actual); Primary Completion 2027-06-04 (Estimated); Study Completion 2027-07-19 (Estimated)

PRIMARY OUTCOMES:
Dual-task walking speed assessment | 6 weeks after subacute stroke
  Speed (m/s)
  The dual-task walking speed assessment measures how well a person walks while simultaneously performing a cognitive or motor task. It helps identify changes in gait speed and stability when attention is divided, revealing potential fall risk or cognitive-motor interference.

SECONDARY OUTCOMES:
Gait Speed assessment | 3 to 6 monts after subacute stroke
  Gait speed (m/s)
Average step duration evaluation | 3 to 6 monts after subacute stroke
  Average step duration (s)
Gait symmetry evaluation | 3 to 6 monts after subacute stroke
  Gait symmetry (%)
Cycle duration variability evaluation | 3 to 6 monts after subacute stroke
  Cycle duration variability (%)
Single-task and double-task gait speed evaluation | 3 to 6 monts after subacute stroke
  Single-task and double-task gait speed difference (%)
Center of pressure position evaluation | up to 6 weeks after subacute stroke
  Lateral variance of center of pressure position (cm²): under two conditions, eyes open and closed.
Proprioception parameters evaluation using Romberg's quotient | up to 6 weeks after subacute stroke
  Romberg's quotient (cm²) The Romberg's quotient is used to evaluate proprioceptive contribution to balance by comparing postural sway with eyes closed versus eyes open.
  It is calculated as:
  Romberg's quotient = Sway with eyes closed / Sway with eyes open A higher quotient suggests greater reliance on visual input for balance and may indicate proprioceptive deficits. This assessment helps determine how well an individual uses proprioception when visual cues are removed.
Balance evaluation using CTSIB-M test | up to 6 weeks after subacute stroke
  Time (s) maintained in CTSIB-M test (s)
  The CTSIB-M (Modified Clinical Test of Sensory Interaction in Balance) assesses a person's ability to maintain balance under four conditions that challenge visual, vestibular, and somatosensory systems. It involves standing on firm and foam surfaces with eyes open or closed, and each condition is timed for up to 30 seconds.
Proprioception using Join Position Sense of the knee test | up to 6 weeks after subacute stroke
  Join Position Sense (°) of the knee. The test involves passively or actively moving the knee to a target angle (e.g., 30° or 60° flexion), then asking the person to replicate that position with eyes closed. The error (in degrees) between the target and reproduced angle reflects proprioceptive precision.

CONTACTS AND LOCATIONS:
Overall Officials: Pauline AMSTUTZ, Principal Investigator — CHR Metz Thionville Hopital Legouest
Locations (1):
- CHR Metz-Thionville Hopital Legouest, Metz, France

IPD SHARING:
Plan to Share IPD: No